CLINICAL TRIAL: NCT01640743
Title: Effect of Different Therapeutic Strategies on Regulatory T Cells in Kidney Transplantation: a Randomized Study
Brief Title: Effect of Different Therapeutic Strategies on Regulatory T Cells in Kidney Transplantation
Acronym: EVERTWIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Carmelo Libetta, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 42501/2009; IRCCS Policlinico S. Matteo (Other: IRCCS Policlinico S. Matteo)
Record Dates: First submitted 2012-07-12; First posted 2012-07-16 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Kidney Transplantation
Keywords: Kidney transplantation; Regulatory T cells; Tolerance; Tacrolimus; Rejection
MeSH Terms: conditions — Rejection, Psychology | interventions — Tacrolimus; Methylprednisolone; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Evertwist 1 (Experimental): Tacrolimus (10-14 ng/ml) + Methylprednisolone (16 mg).
  Interventions: Drug: Tacrolimus + Methylprednisolone
- Evertwist 2 (Experimental): Tacrolimus (4-6 ng/ml) + Everolimus (8-10 ng/ml) + Methylprednisolone (8 mg).
  Interventions: Drug: Tacrolimus + Everolimus + Methylprednisolone

INTERVENTIONS:
Drug: Tacrolimus + Methylprednisolone — Induction therapy:
  Methylprednisolone (500 mg), thymoglobulins (1.5 mg/Kg/die, beginning 1 hour before transplantation) and 1 mg/Kg/die during the following 3 days.
  Maintenance therapy:
  Tacrolimus dosage will be 0.2 mg/kg of body weight and will be administered approximately 12 hours after chirurgical intervention twice a day (mornings and evenings). Dosage will be adapted on individual basis in order to gain pre-dose blood dosages according to indicated plasmatic levels
  Arms: Evertwist 1
Drug: Tacrolimus + Everolimus + Methylprednisolone — Induction therapy:
  Methylprednisolone (500 mg), thymoglobulins (2.5 mg/Kg/die, beginning 1 hour before transplant) and Mycophenolate mofetil (1000 mg) and no immunosuppressive therapy for the following 3 days (WOFIE hypothesis), and for day 4-5-6 thymoglobulins (1.0 mg/Kg/die).
  Maintenance therapy:
  Tacrolimus dosage will be 0.1 mg/kg of body weight and will be administered approximately 12 hours after chirurgical intervention twice a day (mornings and evenings). Dosage will be adapted on individual basis in order to gain pre-dose blood dosages according to indicated plasmatic levels
  Arms: Evertwist 2

SUMMARY:
The objective of the study will be to evaluate the effect of different therapeutic immunosuppressive strategies currently employed in common clinical practice on regulatory T lymphocytes and to verify the hypothesis that the association of thymoglobulins - mTOR inhibitors - small doses of Tacrolimus not only represents a safe anti-rejection therapy but it can also lead to mid-term formation of a high amount of regulatory T cells and, consequently, a high grade of tolerance.

DETAILED DESCRIPTION:
Immune response is mediated by the interaction between antigen-presenting cells (APC), CD4+ helper T cells (Th) and regulatory T cells (Treg), a subpopulation of CD4+ T cells which intensively expresses IL-2 receptor (CD25) and FoxP3 transcription factor. Treg cells contribute maintaining tolerance by suppressing immune response to normal or tumour self-antigens. Treg cells originate in the thymus during ontogenesis and represent approximately 10% of peripheral CD4+ cells. All effector T lymphocytes generate in the thymus at the early stages of life and evolve through the production of new T lymphocytes as well as through antigen-induced expansion of virgin (naive) peripheral T lymphocytes which convert to "memory" T lymphocytes and lie in peripheral lymphoid organs (17). Mature T lymphocytes constitute 70-80% of normal peripheral blood lymphocytes, 30-40% of lymph nodes cells and 20-30% of splenic lymphoid cells.

T lymphocytes are primary effectors of cell-mediated immunity and differentiate into a subpopulation of CD8+ cytotoxic T lymphocytes which are able to lyse foreign cells or virus infected host-cells and a subpopulation of CD4+ T lymphocytes with a regulating activity on T and B lymphocytes and monocytes, through the production of cytokines and cell-to-cell contact.

Treg lymphocytes play a central role among CD4+ cells in balancing tolerance and immunity, as they are responsible for maintaining peripheral tolerance through the control of self-reactive T cells which escaped thymic deletion (19). Studies have in fact demonstrated that whether on one side a defect in their development or activity can lead to serious autoimmune diseases, an excessive immunosuppression mediated by these cells stimulates, on the other side, an immunodeficient condition also towards antigens produced by neoplastic cells favouring, as a consequence, tumour growth.

Treg lymphocytes represent approximately 10% of all CD4+ T cells present in the thymus, peripheral blood and lymphoid tissues; they consist of various populations which differ in terms of particular cell-surface molecules expression and the production of diverse cytokines, but share a common scarce response to antigenic stimulation and an immunosuppressive activity.

The best characterized Treg lymphocytes are the so called "natural occurring Tregs" (nTregs), a sub-group of CD4+ T cells which originates and develops in the thymus during T-cellular maturation process and is afterwards normally present in peripheral blood with the function of controlling self-antigens and preventing autoimmune diseases. These lymphocytes are characterized by the constitutive expression of CD-25 (interleukin-2 receptor α chain), Foxp3 transcription factor (specific to these cells and implied in the development control within the thymus), CTLA-4, GITR and LAG-3 surface molecules as well as TGF-β cytokine, which is present in great quantity on cellular surface and is fundamental to their functioning.

So called "induced Tregs" (iTregs) build the other Treg lymphocytes category: these are CD4+ T lymphocytes which lack in intrinsic regulatory potential but acquire their suppressive activity thanks to a specific and cytokine-mediated activation (26). They are produced in periphery and allow the development of peripheral tolerance to self-antigens, not or scarcely expressed in the thymus. iTregs consist themselves of two different lymphocytic subpopulations: Tr1, present in intestinal mucosa and characterized by a high production of IL-10 and TGF-β but Foxp3 negative; and T helper 3 (Th3), deriving from the induction of native CD4+ T cells due to the ingestion of alimentary antigens, responsible for oral tolerance. Th3 are Foxp3 positive and release high levels of TGF-β (27).

While iTregs seem to function only by the production of immunosuppressive cytokines such as IL-10 and TGF-β, nTregs can exert their activity also through various mechanisms, such as cytokine-dependent, cell contact-dependent or both, according to the nature and intensity of the inflammatory response and of the target tissue to which the latter is directed. This context-dependent regulatory mechanism leads to the elaboration of the model of adaptability and diversification within the function of these cells: in other words, Tregs would constitute a functionally homogeneous cellular subgroup in which every single cell can exert a different mechanism according to the characteristics of inflammatory response. Some authors believe instead that Tregs consist of several subpopulations, each of these presenting its own inhibitory mechanisms (27-28).

Phenotypic characterization of Tregs among circulating human lymphocytes has been complicated by the fact that CD25 is not exclusively expressed by Tregs but also by non-regulatory lymphocytes after activation, so at present only CD4+ cells expressing the highest CD25 levels (CD4+CD25+bright) can be considered authentic Tregs.

In 2003 the Forkhead Transcription Factor (Foxp3) was identified as major regulator in Tregs development; its expression is predominantly restricted to CD4+CD25+ T lymphocytes and Foxp3 expression in naive T cells supports their conversion into a regulatory T phenotype functionally similar to nTregs. Foxp3 is therefore considered an extremely specific marker of Treg cells and is fundamental to the control of their development und functioning. Particularly, some studies have demonstrated that the lack of Foxp3 at birth in humans and rats leads to a massive T-cellular hyperproliferation, resulting in multi-organ autoimmunity and premature death (24), whereas its deletion in adult rats causes hyperproliferation and expansion of dendritic cells as well as death within two weeks. Based on these results Foxp3 seems to be the ideal marker for tolerance study.

Tregs production is strictly controlled by signals emanated by various types of cells, such as epithelial cells, T lymphocytes and APCs. Although the presence of the latter is fundamental to TCR-mediated activation of Tregs, the real suppressive phase in vitro induced by nTregs is actually APC-independent. It implies in fact a mechanism of contact between CD4+CD25- effector T lymphocytes and CD4+CD25+ nTregs.

At present we dispose of little knowledge regarding functional consequences of suppression carried out by Tregs on CD4+ and CD8+ lymphocytes which are sensitive to them, beside that they inhibit IL-2 transcription and, consequently, induce cell cycle interruption. Further immune suppression mechanisms reported by other studies, but not yet confirmed, are following: anergy induction in responsive T cells, refractory reaction to the mitogenic effects of IL-2, release of new iTregs which are likely to suppress Th1s and Th2s by producing TGFβ1 and/or IL-10.

NTregs require particular cytokines for their development and homeostasis. Moreover, Tregs result to be hypoproliferative or anergic to TCR activation, probably due to their incapability of transcribing and actively secreting IL-2. This cytokine is principally released by activated T lymphocytes but not by nTregs and it exerts its biologic activities by binding to its receptor, a membrane protein complex formed by three subunits: α (CD25), β and γ chain.

When IL-2 binds to its receptor in T cells it activates Janus kinases (JAKs) which consequently phosphorylate and release STAT5 proteins (signal transducers and transcription activators). IL-2 exerts in fact its effects on T cells by regulating several target genes primarily at transcriptional level; it does not only increase the expression of IL-2R α and β chains but it also modulates the expression of genes involved in cell cycle regulation, by inducing for instance the up-regulation of proto-oncogenes such as c-myc, c-fos and c-jun, as well as anti-apoptotic genes such as bcl-2 or pro-apoptotic genes like Fas ligand. IL-2 is essential for nTreg development and maintenance, as some studies have demonstrated: induced IL-2 depletion in rats causes autoimmune diseases which can be associated to a reduced number of Foxp3+ nTreg lymphocytes in peripheral compartment.

Another important cytokine to the functioning of Tregs is TGF-β. Despite its inhibitory effects on other T cells, this growth factor is likely to support extra-thymic production of Treg cells and the increase of Foxp3 expression: this action is, however, necessary exclusively to the initial induction. TGF-β plays therefore a different but complementary role to IL-2.

Finally, a further critical cytokine to the functioning of Tr1 lymphocytes is IL-10. Chronic activation in vitro of CD4+ lymphocytes in the presence of IL-10 leads to their differentiation in Tr1, high levels of IL-10 and TGF-β, low levels of IL-2 and IL-4 and a scarce proliferation after restimulation. IL-10 can moreover induce immunosuppression by supporting the formation of anergic T cells capable of inhibiting the activity of other activated T lymphocytes through a contact-dependent mechanism, by competing with the latter for specific APC (Antigen Presenting Cells) receptors and for locally produced IL-2. These anergic T cells are able to suppress immune response in vivo, as their transfer in rats which underwent allogeneic skin graft showed a longer transplant survival.

Beside the above mentioned cytokines, others seem to be involved in different ways in Treg generation and induction, such as IL-4 and IL-13, whereas other cytokines have an antagonist effect on them, such as IL-6 for instance, which contrasts their immunosuppressive activity without interfering with proliferation. Other studies on Treg function have also showed that a transfusion of allogeneic Treg lymphocytes and the subsequent skin graft in IL2Rβ-/- rats (rapidly prone to lethal autoimmune diseases if not treated) not only controlled and suppressed those diseases although Tregs and self-reactive T cells were MHC-incompatible, but also consequently allowed to establish a state of tolerance to those transplants presenting common MHC molecules to donor Tregs. This experiment has then proved that Tregs suppress also self-reactive T cells deriving from non MHC-correlated donors and so, theoretically, that the donor pool for Treg-based immune therapy would be potentially very wide.

Thanks to their essential role in immune tolerance and their immunosuppressive function, Treg lymphocytes are therefore gaining more and more importance in transplantology, as experimental models of organ transplants have underlined their capability of modulating CD4+ and CD8+ cell activity, both responsible for rejection, by inhibiting it, and of suppressing GVHD (Graft-versus-host disease), mediating in this way allotransplant tolerance. There are, however, controversial results regarding Treg phenotype and their action mechanism, depending on the experimental model and on the protocol used to induce this tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged from 18 to 75 years
* Transplanted patients from cadaveric donors
* Patients who has given written informed consensus

Exclusion Criteria:

* Legally unable patients
* Patients who have been participated to others studies in the last 3 months
* Addicted to alcohol or smoking

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2010-03; Primary Completion 2013-06 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Effect of different treatments on absolute and percentual number of regulatory T cells | 12 months
  Comparison of absolute and percentual number of high Treg and FoxP3+ Treg cells in one year post-transplant patients under treatment with different immunosuppressive therapies.

SECONDARY OUTCOMES:
Influence of Treg cell number on renal function and incidence of rejection, death, infection events and cardiovascular diseases. | 24 months
  Comparison of absolute and percentual number variation over time of high Treg and FoxP3+ Treg cells two years after transplant in both groups of patients under treatment, evaluating the influence of Treg cell number on renal function and on incidence of rejection, death, infection events and cardiovascular diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Dal Canton, MD, Study Director — Nephrology Unit, Fondazione Policlinico "San Matteo", Pavia- Italy
Locations (1):
- Fondazione Policlinico "San Matteo", Pavia, Italy

REFERENCES:
- [Background] Taber DJ, Weimert NA, Henderson F, Lin A, Bratton CF, Chavin KD, Baliga PK. Long-term efficacy of induction therapy with anti-interleukin-2 receptor antibodies or thymoglobulin compared with no induction therapy in renal transplantation. Transplant Proc. 2008 Dec;40(10):3401-7. doi: 10.1016/j.transproceed.2008.08.130. PMID 19100399
- [Background] Riley JL, June CH, Blazar BR. Human T regulatory cell therapy: take a billion or so and call me in the morning. Immunity. 2009 May;30(5):656-65. doi: 10.1016/j.immuni.2009.04.006. PMID 19464988
- [Background] Anil Kumar MS, Irfan Saeed M, Ranganna K, Malat G, Sustento-Reodica N, Kumar AM, Meyers WC. Comparison of four different immunosuppression protocols without long-term steroid therapy in kidney recipients monitored by surveillance biopsy: five-year outcomes. Transpl Immunol. 2008 Nov;20(1-2):32-42. doi: 10.1016/j.trim.2008.08.005. Epub 2008 Sep 4. PMID 18773960